CLINICAL TRIAL: NCT03522935
Title: Safety and Tolerability of Escalating Doses of Subcutaneous Elafin (Tiprelestat) Injection in Healthy Normal Subjects
Brief Title: Subcutaneous Elafin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roham T. Zamanian (Other)
Collaborators: Duke University (Other); SRI International (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Roham T. Zamanian, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 42336; P01HL108797 (NIH)
Record Dates: First submitted 2018-02-01; First posted 2018-05-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Elafin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Elafin 0.03 mg/kg (Experimental): 5 subjects will be administered with 0.03 mg/kg of Elafin subcutaneously once daily for 7 days.
  Interventions: Drug: Elafin
- Elafin 0.06 mg/kg (Experimental): 5 subjects will be administered with 0.06 mg/kg of Elafin subcutaneously once daily for 7 days.
  Interventions: Drug: Elafin
- Elafin 0.10 mg/kg (Experimental): 5 subjects will be administered with 0.10 mg/kg of Elafin subcutaneously once daily for 7 days.
  Interventions: Drug: Elafin
- Elafin 0.15 mg/kg (Experimental): 5 subjects will be administered with 0.15 mg/kg of Elafin subcutaneously once daily for 7 days.
  Interventions: Drug: Elafin
- Elafin 0.18 mg/kg (Experimental): 5 subjects will be administered with 0.18 mg/kg of Elafin subcutaneously once daily for 7 days.
  Interventions: Drug: Elafin
- Placebo Drug (Placebo Comparator): 5 subjects will be administered with placebo drug subcutaneously once daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elafin — Elafin subcutaneous.
  Other Names: Tiprelestat
  Arms: Elafin 0.03 mg/kg; Elafin 0.06 mg/kg; Elafin 0.10 mg/kg; Elafin 0.15 mg/kg; Elafin 0.18 mg/kg
Drug: Placebo — Placebo subcutaneous.
  Arms: Placebo Drug

SUMMARY:
A multiple-ascending-dose (MAD), randomized, placebo-controlled, blinded trial to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of Elafin in healthy adult subjects. The purpose of this study is to assess Elafin that is being developed for treatment of PAH. Elafin inhibits elastase, an enzyme that is increased in pulmonary hypertension and is a major factor in the development of PAH. Elafin will be administered subcutaneously daily for 7 days in normal healthy subjects followed over a 28 day time period.

DETAILED DESCRIPTION:
There will be a total of up to 30 subjects randomly assigned to 5 groups with 6 subjects in each group. One subject in each group will be assigned to placebo drug and 5 subjects to active drug. Subjects in each group will receive a single daily dose of Elafin/Placebo for total of 7 days. There will be ascending doses across groups. Groups receiving a higher dose will only do so after the previous group has completed dosing (i.e., 7 days). Each subject will be followed over a 28 day time period.

An interim trial analysis will occur after completion of the 2nd cohort in order for the research team to review PK and safety data to determine modification (if needed) of dosing strategy for groups 3-5. The study is also designed to absorb a de-escalation strategy. If the protocol requires a lowering of dose from the initial dosing, a new group will be assigned a low-dose subcutaneous Elafin regimen.

The study will conclude at any dose that produces clinically significant adverse effects and identified as Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible only if all of the following criteria apply:

1. Male or female, 18 - 55 years of age
2. No history or clinically relevant cardiovascular, renal, gastrointestinal, hepatic, metabolic, endocrine, neurological, or psychiatric abnormalities and is in general good health at screening examination.
3. Normal or clinically acceptable ECG
4. Normal blood pressure (systolic: 90 - 140 mmHg; diastolic: 50 - 90 mmHg) and heart rate (45 - 100 bpm)
5. Body mass index of 18.0 - 32.0 (kg/m2)
6. Ability to communicate well with the investigator and to comply with the requirements of the entire study.
7. Informed consent.
8. Females of childbearing potential must use an acceptable form of contraception at time of enrollment (and throughout the duration of study) including, but not limited to the following:

   1. Documentation of surgical sterilization (bilateral tubal ligation, hysterectomy)
   2. Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing on Day -1 and with an FSH level at screening of ≥ 40 mIU/mL
   3. Intrauterine Device (IUD) plus condom plus contraceptive sponge or foam or jelly
   4. Condom plus contraceptive sponge or foam or jelly
   5. Hormonal contraception (combination oral contraceptives, transdermal patch, injectables, implantables, or vaginal ring) *Subject is not of childbearing potential if the following criteria have been met:

   <!-- -->

   1. Hysterectomy > 1 month ago
   2. Bilateral oophorectomy > 1 month ago
   3. 45-50 years old AND LMP ≥ 24 months ago and documented FSH > 40mIU/mL
9. Males must agree to use a barrier method of birth control from 30 days before first study drug administration until 90 days after last study drug administration.

Exclusion criteria:

A subject will not be eligible if any of the following criteria apply:

1. Administration of any investigational drug 45 days prior to study enrollment.
2. Active participation in another interventional clinical trial.
3. Use of any prescription medication within 30 days (with exception to oral contraceptives) or over-the-counter medication (OTC) within 7 days before first study drug administration. Use of OTC medications may be permitted after day 1 visit until end of study with approval of the protocol investigator.
4. Subject performed heavy physical exertion 2 days before eligibility assessment and before admission into clinical research center.
5. Subject consumes more than 500 mL of beer/day or 250 mL of wine/day or 2 glasses of liquor/day.
6. Subject has a history of chronic alcohol or drug abuse within the last 4 weeks.
7. Subject smokes more than 10 cigarettes per day or has done so within 6 months prior to eligibility assessment.
8. Subject has a diet that deviates notably from the "normal" amounts of protein, carbohydrate, and fat, as judged by the investigator (e.g., vegetarians or vegans).
9. Subject consumes more than 600 mg of caffeine/day (200 mL of coffee contain approximately 100 mg of caffeine, 200 mL of black tea approximately 30 mg and 200 mL of soda approximately 20 mg).
10. Subject has donated blood or had a comparable blood loss (>400 mL) within the last 3 months prior to eligibility assessment or anemia defined by hematocrit value less than 30% at screening.
11. Subject has any clinically relevant abnormality in physical examination, vital signs and electrocardiogram (ECG).
12. Serious adverse reaction or hypersensitivity to any drug.
13. Inability to communicate or co-operate due to a language problem, poor mental development or impaired cerebral function.
14. Females who are lactating or at risk of pregnancy.
15. Presence of pain incurred by unknown causes.
16. History of asthma or other respiratory disease.
17. History of neurologic or neuromuscular disease.
18. History of hypotension, hypertension or cardiovascular disease.
19. History of gastrointestinal, hepatic, or renal disease and/or impairment.
20. Positive urine drug screen for drugs with a high potential for abuse and low persistence in the urine.
21. Subject with active or history of malignancy, known Hepatitis B or C, or HIV.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in healthy controls. | 28 day time period
  Safety and tolerability will be determined on the basis of adverse events reported and the severity of adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: AUC0-last | 28 day time period
  AUC0-last: Area under the concentration time-curve to the last concentration above the lower limit of quantitation (after final dose consumed)

OTHER OUTCOMES:
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: Cmax | 28 day time period
  Cmax: Maximum observed concentration
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: Tmax | 28 day time period
  Tmax: Time of maximum observed concentration
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: Ke | 28 day time period
  Ke: Elimination rate constant
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: AUC0-inf | 28 day time period
  AUC0-inf: Area under the concentration time-curve extrapolated to infinit
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: t½ | 28 day time period
  t½: Terminal elimination half-life
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: CL/F | 28 day time period
  CL/F: Apparent total clearance of the drug from plasma after oral administration
Pharmacokinetic/pharmacodynamic (PK/PD) and immunogenicity parameters in blood sample: V/F | 28 day time period
  V/F: Oral volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Roham T Zamanian, MD, Principal Investigator — Stanford University
Locations (1):
- Duke Early Phase Research Unit (DEPRU), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT03522935/ICF_000.pdf